CLINICAL TRIAL: NCT04659434
Title: A Phase II Study of Anti-PD-1 Antibody (Sintilimab) Plus Rituximab, Gemcitabine and Oxaliplatin (R-GemOx) as Second-line Salvage Therapy in Patients With Relapsed/ Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Sintilimab Plus R-GemOx as Second-line Salvage Therapy in Patients With R/R DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qian Wenbin (Other)
Responsible Party: Sponsor-Investigator, Qian Wenbin, Hematology Department Director, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2020001398
Record Dates: First submitted 2020-11-26; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Sintilimab 200mg ivdrip Q3W; Rituximab 375mg/m2 ivdrip; Gemcitabine 1000mg ivdrip; Oxaliplatin 100mg/m2 ivdrip
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Patients receive sintiliman+R-GemOx three weeks for a cycle, detailed as follows:
  Combination therapy
  * Anti-PD-1 antibody (sintilimab): Fixed dose of 200 mg every 3 weeks, d0, intravenous drip (without pretreatment), infusion time: 30 mintutes (no less than 20 mins, no more than 60 mins), for 4 cycles
  * R-GemOx: Rituximab 375mg/m2, d1; Gemcitabine 1000mg, d2; Oxaliplatin 100mg/m2, d2; every 3 weeks for a cycle, 4 cycle as protocol specified.
  Monotherapy:
  -Anti-PD-1 antibody (sintilimab): Fixed dose of 200 mg every 3 weeks, d0, intravenous drip (without pretreatment), infusion time: 30 mintutes (no less than 20 mins, no more than 60 mins), for 8 cycles
  Other Names: IBI308

SUMMARY:
This study evaluates the addition of Sintilimab to current 2nd line salvage therapy of Rituximab, Gemcitabine and Oxaliplatin (R-GemOx) for patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL). All patients will receive four cycles of sintilimab plus R-GemOx. Afterwards, 1) patients who achieve CR assessed by PET-CT and are eligible for autologous stem cell transplantation (ASCT) will undergo ASCT. After transplantation, patients will receive sintilimab monotherapy up to 8 cycles or until disease recurrence and progression, death, intolerance and toxicity, withdrawal of informed consent, or other reasons specified in the protocol. 2) Patients who achieve CR assessed by PET-CT and are not eligible for ASCT will directly receive sintilimab monotherapy as maintenance treatment for a maximum of 8 cycles as described above. 3) Patients achieved PR, SD or PD assessed by PET/CT will withdraw from this study and receive proper treatment based on investigator's decision.

DETAILED DESCRIPTION:
Rituximab is a chimeric mouse/human monoclonal antibody that binds to CD20, on pre-B and mature B lymphocytes and eliminates these cells potentially via a number of different mechanisms. The R-GemOx regimen has been adopted by numerous medical institutions internationally as therapy for older patients or comorbid patients with relapsed or refractory DLBCL and as a back-bone for the investigation of novel therapies in combination with chemotherapy. The cytotoxic T-lymphocyte co-receptor PD-1 has been extensively studied and is recognized to provide critical inhibitory signals that down-regulate T-cell function and provides a mechanism for immune evasion for tumors. PD-L1, the ligand of PD-1 is expressed on DLBCL tumor cells, along with infiltrating non-malignant cells, primarily macrophages, with PD-1 expressed on tumor infiltrating lymphocytes (TILs). Sintilimab targets programmed PD-1 on tumor cells and prevents interaction with either PD-1 receptor or B7.1 (CD80), both of which function as inhibitory receptors expressed on T cells. Interference of the PD-L1:PD-1 and PDL1:B7.1 interactions may enhance the magnitude and quality of the tumor-specific T-cell response through increased T-cell priming, expansion, and/or effector function. This study of sintilimab in combination with rituximab, gemcitabine and oxaliplatin aims to address the unmet clinical need of patients with relapsed and refractory DLBCL. It is based upon a sound mechanistic approach, investigating the activity of novel agents and will aim to compressively explore biomarkers of response. The primary objective will be the complete response rate (CRR) of this salvage therapy. A maintenance phase of sintilimab will be added as this may induce an on-going T-cell response to neo-antigens released as a result of previous treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent.
2. Age range from 18 to 80 years;
3. Pathologically confirmed CD20+ diffuse large B-cell lymphoma
4. According to Lugano 2014, at least one measurable nodular lesion with a length of greater than 15 mm, or extranodal lesion greater than 10 mm, lesion on FDG-PET scan demonstrates uptake);
5. Diffuse large B-cell lymphoma patients failed to first-line rituximab based chemotherapy including anthracycline or anthracycline
6. Patients are allowed to receive palliative radiotherapy, but the last time radiotherapy cannot be within 7 days before the first study drug administration;
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
8. Adequate organ function
9. Expectation survival time over 3 months;

Exclusion Criteria:

1. History of other malignancy within the past 5 years (except for 1. basal cell carcinoma of the skin and 2. carcinoma in situ of the cervix and 3. patients who had received treatment for the purpose of cure and had not developed a malignant tumor with a known active disease in the previous 5 years);
2. Patients who had received other antitumor therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks before the start of the enrollment (if patients received small-molecule targeted drug therapy, they could be included in the study if the drug was discontinued for more than 5 half-lives), or had not recovered from the previous toxicity;
3. Previous treatment with anti-PD-1 antibody, anti-PD-L1 antibody or other medications that stimulates or collaboratively inhibits T cell receptors
4. Patients previously received anti-CD20 antibody combined GemOx regimen;
5. Evidence of central nervous system invasion;
6. Patients received systemic treatment of traditional Chinese herb with anti-tumor indications or immunomodulatory drugs (including thyroxin, interferon and interleukinin, except for local use to control pleural effusions) within 2 weeks before first administration;
7. Patients with autoimmune diseases requiring treatment or with a history of syndrome requiring systemic use of steroid immunosuppressive agents, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc;
8. Patients received systemic glucocorticoid therapy (excluding nasal spray, inhaled or other topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to the first administration;
9. Clinically uncontrollable pleural effusion/peritoneal effusion (patients who do not need drainage effusion or do not significantly increase the effusion after 3 days of drainage can be enrolled);
10. Patients who have had previous organ transplants (except autologous hematopoietic stem cell transplants);
11. Patients are allergic to sintilimab, CD20 monoclonal antibody and GemOx regimen
12. Patients has not fully recovered from toxicity and/or complications due to any intervention prior to initiation of treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss);
13. A confirmed history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
14. A confirmed history of Novel Coronavirus infection;
15. Patients with hepatitis B (HBV HBsAg positive and HBV-DNA≥105), hepatitis C (HCV) infection (HCV antibody positive and HCV-RNA detectable); And subjects with other acquired or congenital immune deficiency diseases, including but not limited to hiv-infected;
16. Patients who received the live vaccine within 4 weeks of the start of the enrollment;
17. Pregnant or lactating women;
18. Patients who have received grade II or above surgery within 3 weeks before enrollment;
19. Patients with significant coagulation abnormality;
20. Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interfere with results interpretation, including uncontrolled diabetes, or pulmonary disease (a history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm);
21. Patients who received the live vaccine within 4 weeks of the start of the enrollment;
22. Severe or uncontrolled infections;
23. Patients with history of severe neurological or psychiatric illness, including dementia or epilepsy;
24. Patients with drug abuse, medical, psychological or social conditions that may interfere with the study results or the assessment of the study results;
25. Patients are unsuitable for the enrollment according to investigator's judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-12-10 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 6 weeks after the last dose of the combination therapy (each cycle is 21 days)
  Complete response rate after treated by Sintilimab and R-GemOx

SECONDARY OUTCOMES:
Over response rate (ORR) | 6 weeks after the last dose of the combination therapy (each cycle is 21 days)
  Overall response rate after treated by Sintilimab and R-GemOx
Overall Survival (OS) | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Rate of grade 3 or 4 treatment related adverse effect | Time Frame: Up to 30 days after the last cycle of per-protocol treatment and 90 days after last dose of anti-PD-1 antibody (each cycle is 28 days)
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: wenbin Qian, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No